CLINICAL TRIAL: NCT01649193
Title: Determining the Minimal Important Difference of the Short Physical Performance Battery and 4m Gait Speed in Chronic Respiratory Disease Patients.
Brief Title: What is an Important Change in the Short Physical Performance Battery (SPPB)?
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2012LF001H
Record Dates: First submitted 2012-07-09; First posted 2012-07-25 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Respiratory Tract Diseases; Lung Diseases
Keywords: Rehabilitation [E02.831]; Exercise [G11.427.394.380]; Health Education [I02.233.332]; [C08]; [C08.381]
MeSH Terms: conditions — Respiratory Tract Diseases; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood taken and stored as whole blood, serum, and plasma.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Respiratory Disease: Any patient with a chronic respiratory disease referred for pulmonary rehabilitation
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation — An eight week out-patient based programme consisting of twice weekly supervised exercise and educational sessions

SUMMARY:
The purpose of this study is to determine the important change in the Short Physical Performance Battery (SPPB) when used in patients with lung disease. The SPPB is a simple physical test that measures balance and the functioning of the legs. It has been widely used in healthy elderly populations and predicts hospital admission and the onset of disability. The SPPB has not previously been used in patients with lung disease, and it is not clear what change in this test is considered meaningful and worthwhile by patients or doctors (the minimal clinically important difference: MID). Knowing what the MID for the SPPB will allow researchers and doctors to evaluate the effectiveness of current and new treatments, and to detect improvement or deterioration in the condition of patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients entering pulmonary rehabilitation

Exclusion Criteria:

* Any patient in whom mobility and lower limb function have been significantly affected by a neuromuscular cause, severe peripheral vascular disease or amputation.
* Any patient whom the chief investigator feels it is unsafe to exercise (e.g. unstable cardiac disease).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All chronic respiratory disease patients referred for pulmonary rehabilitation.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Short Physical Performance Battery | 8 weeks

SECONDARY OUTCOMES:
Change from baseline of MRC Dyspnoea Scale | 8 weeks
Change from baseline of St George's Respiratory Questionaire | 8 weeks
Anchor question (5-point Likert scale) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William DC Man, MRCP, PhD, Principal Investigator — Repiratory Biomedical Reserach Unit, Royal Brompton & Harefield NHS Foundation Trust and Imperial College London
Locations (1):
- Harefield Hospital, Harefield, Middlesex, United Kingdom

REFERENCES:
- [Background] Singh SJ, Morgan MD, Scott S, Walters D, Hardman AE. Development of a shuttle walking test of disability in patients with chronic airways obstruction. Thorax. 1992 Dec;47(12):1019-24. doi: 10.1136/thx.47.12.1019. PMID 1494764
- [Background] Jones PW, Quirk FH, Baveystock CM, Littlejohns P. A self-complete measure of health status for chronic airflow limitation. The St. George's Respiratory Questionnaire. Am Rev Respir Dis. 1992 Jun;145(6):1321-7. doi: 10.1164/ajrccm/145.6.1321. PMID 1595997
- [Background] Guralnik JM, Ferrucci L, Simonsick EM, Salive ME, Wallace RB. Lower-extremity function in persons over the age of 70 years as a predictor of subsequent disability. N Engl J Med. 1995 Mar 2;332(9):556-61. doi: 10.1056/NEJM199503023320902. PMID 7838189
- [Derived] Nolan CM, Kon SSC, Patel S, Jones SE, Barker RE, Polkey MI, Maddocks M, Man WD. Gait speed and pedestrian crossings in COPD. Thorax. 2018 Feb;73(2):191-192. doi: 10.1136/thoraxjnl-2017-210173. Epub 2017 May 5. PMID 28476882